CLINICAL TRIAL: NCT01501305
Title: Influence of Carob and Probiotics on Acute Diarrhea in Children
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 68-2010
Record Dates: First submitted 2011-12-26; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Diarrhea
Keywords: influence; carob powder; probiotics; duration
MeSH Terms: conditions — Diarrhea | interventions — Probiotics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Mineral rehydration solution
  Interventions: Dietary Supplement: Mineral solution
- Carob powder (Active Comparator): Carob powder and probiotics
  Interventions: Dietary Supplement: Carob powder with probiotics

INTERVENTIONS:
Dietary Supplement: Mineral solution — Rehydration mineral solution
  Arms: Placebo
Dietary Supplement: Carob powder with probiotics — 7 1/2 grams of carob powder and probiotic twice daily for one week or until diarrhea is gone
  Arms: Carob powder

SUMMARY:
Comparison of Carob powder with probiotics vs oral hydration solution in diarrhea treatment in children.

ELIGIBILITY:
Inclusion Criteria:

* Acute diarrhea

Exclusion Criteria:

* Dehydration
* Chronic diseases
* Chronic diarrhea (more than 2 weeks)
* Septic shock
* Hypovolemia
* On medication
* Pregnancy

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Reduction in diarrhea | One week
  Measurement of number of vomiting and diarrhea bowel movements before and after intervention

SECONDARY OUTCOMES:
Number of days until no diarrhea bowel movements | 1 week
  Measurement of number of days until diarrhea is gone

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel